CLINICAL TRIAL: NCT00561067
Title: Evaluation of the Tolerability and Efficacy of Erythropoietin (EPO) Treatment in Spinal Shock: Comparative Study VS Methylprednisolone (MP)
Brief Title: Evaluation of Tolerability and Efficacy of Erythropoietin (EPO) Treatment in Spinal Shock: Comparative Study Versus Methylprednisolone (MP)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Italian Medicines Agency decision
Sponsor: Niguarda Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FARM6Y35XM
Record Dates: First submitted 2007-11-19; First posted 2007-11-20 (Estimated); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Spinal Cord Injury
Keywords: Spinal cord injury; spinal shock; erythropoietin
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Erythropoietin; Methylprednisolone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Methylprednisolone
  Interventions: Drug: Methylprednisolone
- 2 (Experimental): Erythropoietin
  Interventions: Drug: Erythropoietin

INTERVENTIONS:
Drug: Erythropoietin — EPO 500 IU/kg diluted in 50 ml saline and infused in 30 minutes; treatment is started within eight hours after the spinal injury; the same drug dosage will be infused at 24 and 48 hours
  Arms: 2
Drug: Methylprednisolone — MP 30 mg/kg intravenous (iv) in the first hour, followed by 5.4 mg/kg/h for 23 hours if treatment is started within three hours after the spinal injury,or for 48 hours if treatment is started between three and eight hours (protocol NASCIS III, National Acute Spinal Cord Injury Study)
  Arms: 1

SUMMARY:
The purpose of this study is to evaluate the tolerability and efficacy of erythropoietin (EPO) treatment in spinal shock in comparison with the methylprednisolone treatment (MP).

DETAILED DESCRIPTION:
Traumatic spinal cord injury (TSCI) is devastating for the patient and costly to society. Currently, methylprednisolone (MP) administered according NASCIS (III) protocol is the only therapy which has minor benefits and is accompanied by dangerous side effects. Any new treatment of TSCI that allows major recovery of function would be a significant advance in clinical care. Much of the motor and sensory paralysis following TSCI occurs because of a delayed and widespread oligodendrocyte apoptosis and demyelination of long spinal tracts. We have recently reported that erythropoietin (EPO) administration significantly attenuates such delayed secondary degeneration and promotes functional recovery in TSCI animal models. The research proposed is a multicenter trial involving the Italian Spinal Units that have developed a multidisciplinary experience on the management of TSCI. Primary objective of the study is to assess the superiority of EPO compared to MP in improving the clinical outcome of SCI (ASIA Impairment Scale); secondary objectives are: to assess the safety of EPO compared to MP, the effects on the motor and sensory functions and on improving functional autonomy, the influence on spasticity and neurogenic pain, and, the impact on surrogate end-points (Somatosensory Evoked Potentials and Magnetic Resonance Imaging).The study population is characterized by all patients with TSCI (ASIA Impairment Scale A or B) admitted to Italian Spinal Units: we estimate an enrolment of 100 subjects , 50 in each therapeutic arm. The study proposed is a single-blind randomized phase III parallel group trial in which eligible patients are randomized to one of the following treatment modalities: MP according to NASCIS III protocol or EPO iv (500 UI/kg within 8 hours after the SCI, dosage repeated at 24 and 48 hours). The duration of the study will be 24 months, with a 21-month maximum time to engage all the patients required by the power calculation.The primary end-point will be assessed using the Cochrane-Mantel-Haenzel test; the changes in the SEP (latency) and size of the MRI lesions using the Repeated Measures Analysis of Variance (ANOVA), the Ashworth, VAS, PENN, and SCIM scores with the parametric Wilcoxon's signed-ranks test. The effect of treatment on the primary end-point will be evaluated using a multivariate analysis model (binary logistic regression). The non-parametric alternative will be conducted if the assumption of normality will be not verified.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic SCI occurred within 8 hours
* Hemodynamic stability at the time of treatment start (systolic blood pressure > 90 mmHg for at least 1 hour without massive infusion or vasopressor support for ongoing bleeding)
* Neurological level between C5 and T12 (ASIA scale)
* ASIA Impairment Scale: A or B
* Informed consent

Exclusion Criteria:

* SCI other than traumatic
* SCI caused by edged weapons or fire arms
* Traumatic SCI after 8 hours
* Neurological level above C5 or below T12
* ASIA Impairment Scale C, D, E
* Uncontrolled arterial hypertension
* Past or current cerebrovascular disease
* Past or current acute myocardial infarction
* History of thrombotic events
* Other chronic cardiovascular disorders (cardiac arrhythmias, congestive heart failure)
* History of peripheral arterial disease, polycythemia, porphyria, active malignancy
* Previous or current neurological diseases with abnormal neurological examination
* Suspected or definite pregnancy or lactation (requiring ßHCG confirmation)
* Clinically relevant psychiatric disease
* Known allergy to EPO
* Hypersensitivity to human albumin
* Acute or chronic renal failure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-04 (Actual); Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Improvement of ASIA Impairment Scale of at least 1 grade. Score on ASIA Scale and a ASIA Impairment Scale are an inclusion criteria, then at 3rd, 7th, 14th, 30th, 60th, 90th days | 3 months

SECONDARY OUTCOMES:
Increase of ASIA motor/sensory scores at 3rd, 7th, 14th, 30th, 60th, 90th days | 3 months
Functional autonomy with SCIM scores at 7th, 30th, 60th, 90th days | 3 months
Spasticity with the Ashworth Scale, spasms with the PENN Scale and neurogenic pain with the VAS Scale at 7th, 14th days | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Tiziana Redaelli, MD, Principal Investigator — Azienda Ospedaliera Ospedale Niguarda Ca' Granda Milano
Locations (1):
- A.O. Ospedale Ca' Granda, Milan, Italy